CLINICAL TRIAL: NCT01065688
Title: A Prospective Randomized Controlled Trial Comparing Billroth-I Reconstruction With Roux-en Y Reconstruction After Distal Gastrectomy for Gastric Cancer
Brief Title: A Trial of Reconstruction After Distal Gastrectomy for Gastric Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Wakayama Medical University (Other)
Responsible Party: Principal Investigator, Hiroki Yamaue, Second Department of Surgery, Wakayama Medical University, Wakayama Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: WMU-GC03
Record Dates: First submitted 2010-02-08; First posted 2010-02-09 (Estimated); Last update posted 2018-10-09 (Actual); Status verified 2018-10

CONDITIONS: Gastric Cancer
Keywords: distal gastrectomy; Billroth-I reconstruction; gastric cancer; QOL
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Roux-en Y (Active Comparator): Roux-en Y reconstruction after distal gastrectomy
  Interventions: Procedure: Roux-en Y reconstruction
- Billroth-I (Experimental): Billroth-I reconstruction after distal gastrectomy
  Interventions: Procedure: Billroth-I reconstruction

INTERVENTIONS:
Procedure: Roux-en Y reconstruction — surgical procedure
  Arms: Roux-en Y
Procedure: Billroth-I reconstruction — surgical procedure
  Arms: Billroth-I

SUMMARY:
The purpose of this study is to evaluate the quality of life (QOL) after Billroth-I reconstruction (B-I) following distal gastrectomy, compared with Roux-en Y reconstruction (R-Y) in patients with gastric cancer.

DETAILED DESCRIPTION:
The purpose of this study is to evaluate the quality of life (QOL) after Billroth-I reconstruction (B-I) following distal gastrectomy, compared with Roux-en Y reconstruction (R-Y) in patients with gastric cancer. There is no prospective randomized study of the two operative procedures focusing on postoperative QOL. The investigators conducted a prospective randomized trial on 120 patients who underwent distal gastrectomy comparing Billroth-I reconstruction and Roux-en Y reconstruction.

The primary endpoint was the postoperative QOL. The secondary endpoints were the incidence of postoperative complications, nutritional status, and the incidence of the remnant gastritis and the reflux esophagitis. Patients were recruited into this study before surgery, on the basis of whether distal gastrectomy was anticipated at Wakayama Medical University Hospital(WMUH) for gastric cancer, and appropriate informed consent was obtained. Exclusion criteria was 1) patients with severe complications which were possible to prolong hospital stay, 2) patients with history of other organ malignancies, 3) patients who were diagnosed inadequacy for this study by a physician, and 4) patients without an informed consent.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed adenocarcinoma of stomach
* Performance status: Eastern Cooperative Oncology Group (ECOG) 0-1
* Tumor located in the antrum or the angle or the lower body of stomach
* Appropriate informed consent was obtained.

Exclusion Criteria:

* Patients with severe complications which were possible to prolong hospital stay
* Patients with history of other organ malignancies
* Patients who were diagnosed inadequacy for this study by a physician
* Patients without an informed consent

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2009-01; Primary Completion 2013-09 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
the postoperative quality of life (QOL) | 3 years after operation

SECONDARY OUTCOMES:
the incidence of postoperative complications, nutritional status, and the incidence of the remnant gastritis and the reflux esophagitis | 1, 3 and 5 years after operation

CONTACTS AND LOCATIONS:
Overall Officials: Masaki Nakamura, MD, Principal Investigator — Second Department of Surgery, Wakayama Medical University
Locations (1):
- Second Department of Surgery, Wakayama Medical University, Wakayama, Japan

REFERENCES:
- [Background] Ojima T, Iwahashi M, Nakamori M, Nakamura M, Naka T, Katsuda M, Iida T, Tsuji T, Hayata K, Takifuji K, Yamaue H. Clinicopathological characteristics of remnant gastric cancer after a distal gastrectomy. J Gastrointest Surg. 2010 Feb;14(2):277-81. doi: 10.1007/s11605-009-1090-5. PMID 19911236
- [Background] Ojima T, Iwahashi M, Nakamori M, Nakamura M, Naka T, Katsuda M, Iida T, Hayata K, Yamaue H. Association of allogeneic blood transfusions and long-term survival of patients with gastric cancer after curative gastrectomy. J Gastrointest Surg. 2009 Oct;13(10):1821-30. doi: 10.1007/s11605-009-0973-9. Epub 2009 Aug 5. PMID 19655208
- [Background] Iwahashi M, Nakamori M, Nakamura M, Naka T, Ojima T, Iida T, Katsuda M, Ueda K, Yamaue H. Evaluation of double tract reconstruction after total gastrectomy in patients with gastric cancer: prospective randomized controlled trial. World J Surg. 2009 Sep;33(9):1882-8. doi: 10.1007/s00268-009-0109-0. PMID 19548028
- [Background] Ojima T, Iwahashi M, Nakamori M, Nakamura M, Naka T, Ishida K, Ueda K, Katsuda M, Iida T, Tsuji T, Yamaue H. Influence of overweight on patients with gastric cancer after undergoing curative gastrectomy: an analysis of 689 consecutive cases managed by a single center. Arch Surg. 2009 Apr;144(4):351-8; discussion 358. doi: 10.1001/archsurg.2009.20. PMID 19380649
- [Derived] Nishizaki D, Ganeko R, Hoshino N, Hida K, Obama K, Furukawa TA, Sakai Y, Watanabe N. Roux-en-Y versus Billroth-I reconstruction after distal gastrectomy for gastric cancer. Cochrane Database Syst Rev. 2021 Sep 15;9(9):CD012998. doi: 10.1002/14651858.CD012998.pub2. PMID 34523717
- [Derived] Nakamura M, Nakamori M, Ojima T, Iwahashi M, Horiuchi T, Kobayashi Y, Yamade N, Shimada K, Oka M, Yamaue H. Randomized clinical trial comparing long-term quality of life for Billroth I versus Roux-en-Y reconstruction after distal gastrectomy for gastric cancer. Br J Surg. 2016 Mar;103(4):337-47. doi: 10.1002/bjs.10060. Epub 2016 Feb 3. PMID 26840944